CLINICAL TRIAL: NCT05492552
Title: Cardiovascular Implications and Physical Activity in Middle-age and Older People With a History of Coronavirus 2019 (COVID-19)
Brief Title: Cardiovascular Function and Physical Activity in COVID-19
Acronym: CV-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Responsible Party: Principal Investigator, Djordje Jakovljevic, Principle Investigator, Coventry University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P125303
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Coronavirus 2019
Keywords: Coronavirus 2019; Cardiovascular System; Arterial Stiffness; Echocardiography; Cardiopulmonary exercise stress testing; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-COVID participants (No Intervention)
- COVID participants in intervention (Experimental): The intervention group will attend the laboratory for baseline testing and complete a week of usual daily activity. Following this week they will then be guided to increase their daily step count by 2,000 and supported through weekly telephone calls.
  Interventions: Behavioral: Active-at-home-HF
- COVID participants assigned to usual daily activity (No Intervention)

INTERVENTIONS:
Behavioral: Active-at-home-HF — Increase daily step count by 2,000 and weekly telephone calls.
  Arms: COVID participants in intervention

SUMMARY:
The purpose of this study is to a) assess how coronavirus 2019 (COVID-19) affects cardiac function in middle age and older adults and b) assess if a physical activity intervention (increased daily step count by 2,000) can affect cardiac function in a population with a history of COVID-19.

DETAILED DESCRIPTION:
Cardiac function will be assessed by obtaining arterial stiffness, comprehensive echocardiography measurements and haemodynamic monitoring. Arterial stiffness will assess primarily pulse wave velocity (PWV) and echocardiography. Graded cardiopulmonary exercise stress testing coupled with non-invasive gas exchange and haemodynamic monitoring will also be performed. Physical activity will be assessed objectively using pedometers and accelerometry. Quality of life, sleep/ circadian rhythm, fatigue, anxiety and depression will be measured using the validated Short-Form-36 (SF-36) questionnaire, Pittsburgh Sleep scale (PSQI), Chalder fatigue (CF) scale and the Depression, Anxiety and Stress Scale (DASS-21).

ELIGIBILITY:
Inclusion Criteria:

* Between 50-85 years old
* Up to date with all COVID-19 vaccinations
* COVID participants - had a positive test for COVID-19 over 28 days of initial visit but before 18 months. Non-COVID participants - never received a positive COVID-19 test result, and no symptoms during periods where testing was unavailable.

Exclusion Criteria:

* Chronic respiratory and cardiovascular conditions i.e., chronic obstructive pulmonary disease (COPD), emphysema, pulmonary hypertension, coronary artery disease
* Severe hypertension
* Acute or chronic neurological impairment or progressive neurological disease
* Use of medication known to directly affect cardiac function
* Current smoker
* Body mass index > 35 kg/m2
* People who exceed current physical activity guidelines defined by the World Health Organization (WHO).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Difference and change in left ventricular global longitudinal strain. | 12 weeks (baseline to 12 weeks)
  1. Difference in left ventricular global longitudinal strain between COVID and non-COVID participants at rest and during peak exercise on baseline assessment.
  2. Change in left ventricular global longitudinal strain between COVID intervention and COVID usual care group at rest and during peak exercise on baseline and end of study assessments.
  Left ventricular global longitudinal strain is measured as a percentage (%) using transthoracic echocardiography.

SECONDARY OUTCOMES:
Difference and change in pulse wave velocity. | 12 weeks (baseline to 12 weeks)
  1. Difference in pulse wave velocity between COVID and non-COVID participants at baseline assessment.
  2. Change in pulse wave velocity between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Pulse wave velocity (a measure of arterial stiffness) will be measured in meters per second (m/s) using a tonometer and sphygmomanometer.
Difference and change in augmentation index. | 12 weeks (baseline to 12 weeks)
  1. Difference in augmentation index between COVID and non-COVID participants at baseline assessment.
  2. Change in augmentation index between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Augmentation index (a measure of arterial stiffness) will be measured as percentage (%) using sphygmomanometer.
Difference and change in resting cardiac output. | 12 weeks (baseline to 12 weeks)
  1. Difference in resting cardiac output between COVID and non-COVID participants at baseline assessment.
  2. Change in resting cardiac output between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Cardiac output (i.e. volume of blood ejected from the heart) will be measured in litres per minute (L/min) using non-invasive monitoring technology.
Difference and change in maximal cardiac output. | 12 weeks (baseline to 12 weeks)
  1. Difference in maximal cardiac output between COVID and non-COVID participants at baseline assessment.
  2. Change in maximal cardiac output between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Cardiac output (i.e. volume of blood ejected from the heart) will be measured in litres per minute (L/min) using non-invasive monitoring technology.
Difference and change in resting heart rate. | 12 weeks (baseline to 12 weeks)
  1. Difference in resting heart rate between COVID and non-COVID participants at baseline assessment.
  2. Change in resting heart rate between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Heart rate (i.e. times the heart beats per minute) will be measured using non-invasive monitoring technology.
Difference and change in maximal heart rate. | 12 weeks (baseline to 12 weeks)
  1. Difference in maximal heart rate between COVID and non-COVID participants at baseline assessment.
  2. Change in maximal heart rate between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Heart rate (i.e. times the heart beats per minute) will be measured using non-invasive monitoring technology.
Difference and change in resting stroke volume. | 12 weeks (baseline to 12 weeks)
  1. Difference in resting stroke volume between COVID and non-COVID participants at baseline assessment.
  2. Change in resting stroke volume between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Stroke volume (i.e. volume of blood pumped out of the heart in one beat) will be measured in liters (L) using non-invasive monitoring technology.
Difference and change in maximal stroke volume. | 12 weeks (baseline to 12 weeks)
  1. Difference in maximal stroke volume between COVID and non-COVID participants at baseline assessment.
  2. Change in maximal stroke volume between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Stroke volume (i.e. volume of blood pumped out of the heart in one beat) will be measured in liters (L) using non-invasive monitoring technology.
Difference and change in resting systemic vascular resistance. | 12 weeks (baseline to 12 weeks)
  1. Difference in resting systemic vascular resistance between COVID and non-COVID participants at baseline assessment.
  2. Change in resting systemic vascular resistance between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Systemic vascular resistance (i.e. the force exerted on circulating blood by the vasculature of the body) will be measured in mmHg⋅min/mL using non-invasive monitoring technology.
Difference and change in maximal systemic vascular resistance. | 12 weeks (baseline to 12 weeks)
  1. Difference in maximal systemic vascular resistance between COVID and non-COVID participants at baseline assessment.
  2. Change in maximal systemic vascular resistance between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Systemic vascular resistance (i.e. the force exerted on circulating blood by the vasculature of the body) will be measured in mmHg⋅min/mL using non-invasive monitoring technology.
Difference and change in maximal oxygen uptake (VO2 max). | 12 weeks (baseline to 12 weeks)
  1. Difference in VO2 max between COVID and non-COVID participants at baseline assessment.
  2. Change in VO2 max between COVID intervention and COVID usual care group at baseline and end of study assessments.
  VO2 max (i.e. maximal oxygen uptake) will be measured in milliliters per minute (mL/min).
Difference and change in Forced Expiratory Volume 1 (FEV1)/ forced vital capacity (FVC) ratio. | 12 weeks (baseline to 12 weeks)
  1. Difference in FEV/FEV1 ratio between COVID and non-COVID participants at baseline assessment.
  2. Change in FEV/FEV1 ratio between COVID intervention and COVID usual care group at baseline and end of study assessments.
  FEV/FEV1 ratio (i.e. the ratio that reflects the amount of air you can forcefully exhale from your lungs) will be measured using spirometry.
Change in quality of life measured by the SF-36 questionnaire between baseline and post intervention assessment at 12 weeks. | 12 weeks (baseline to 12 weeks)
  Difference in quality of life 36 Item Short Form survey scores between baseline and end of study assessments.Score ranges from 0-100, with higher scores associated with a better outcome.
Difference and change in depression, anxiety and stress measured on the DASS-21 questionnaire. | 12 weeks (baseline to 12 weeks)
  1. Difference in depression, anxiety and stress between COVID and non-COVID participants at baseline assessment.
  2. Change in depression, anxiety and stress between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Depression, anxiety and stress measured on the DASS-21 questionnaire. Score ranges from 0-56, with higher scores associated with a worse outcome.
Difference and change in global sleep efficiency. | 12 weeks (baseline to 12 weeks)
  1. Difference in global sleep efficiency between COVID and non-COVID participants at baseline assessment.
  2. Change in global sleep efficiency between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Sleep efficiency is measured on the Pittsburgh Sleep Quality Index (PSQI) questionnaire. Score ranges from 0-21, with higher scores associated with a worse outcome.
Change in sleep efficiency. | 12 weeks (baseline to 12 weeks)
  1. Difference in sleep efficiency between COVID and non-COVID participants at baseline assessment.
  2. Change in sleep efficiency between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Sleep efficiency is measured using the Condor Actigraph watch. Score ranges from 0-100%, with higher scores associated with a higher sleep efficiency.
Difference and change in right ventricular global longitudinal strain. | 12 weeks (baseline to 12 weeks)
  1. Difference in resting right ventricular global longitudinal strain between COVID and non-COVID participants at baseline assessment.
  2. Change in resting right ventricular global longitudinal strain between COVID intervention and COVID usual care group at baseline and end of study assessments.
  Right ventricular global longitudinal strain is measured as a percentage (%) using transthoracic echocardiography.
Difference and change in left atrial strain. | 12 weeks (baseline to 12 weeks)
  1. Difference in left atrial strain between COVID and non-COVID participants at rest and during exercise on baseline assessment.
  2. Change in left atrial strain between COVID intervention and COVID usual care group at rest and during exercise on baseline and end of study assessments.
  Left atrial strain is measured as a percentage (%) using transthoracic echocardiography.
Difference and change in ventricular arterial coupling. | 12 weeks (baseline to 12 weeks)
  1. Difference in ventricular arterial coupling between COVID and non-COVID participants on baseline assessment.
  2. Change in ventricular arterial coupling between COVID intervention and COVID usual care group on baseline and end of study assessments.
  Ventricular arterial coupling (VAC) is a ratio which is calculated using the formula VAC = Ea/Ees; where Ea = arterial elastance (0.9 x systolic blood pressure/ stroke volume) and Ees = ventricular elastance (0.9 x systolic blood pressure/ left ventricular end systolic volume (LVESV).
  stroke volume and LVESV are both calculated using echocardiography techniques.
Difference and change in right ventricular diastolic function. | 12 weeks (baseline to 12 weeks)
  1. Difference in right ventricular diastolic function between COVID and non-COVID participants on baseline assessment.
  2. Change in right ventricular diastolic function between COVID intervention and COVID usual care group on baseline and end of study assessments.
  Right ventricular diastolic function has no particular units, rather is graded impaired or restrictive right ventricular filling using several echocardiographic measurements i.e., tricuspid valve E:A ratio, tricuspid valve deceleration time (milliseconds (ms)).
Difference and change in electrocardiography (ECG) R-R interval average. | 12 weeks (baseline to 12 weeks)
  1. Difference in R-R average between COVID and non-COVID participants at rest on baseline assessment.
  2. Change in R-R average between COVID intervention and COVID usual care group at rest on baseline and end of study assessments.
  R-R average is a measurement of Heart Rate Variability, measured in milliseconds (ms) using electrocardiography.
Difference and change in root mean square of successive ECG RR interval difference (RMSSD). | 12 weeks (baseline to 12 weeks)
  1. Difference in RMSSD between COVID and non-COVID participants at rest on baseline assessment.
  2. Change in RMSSD between COVID intervention and COVID usual care group at rest on baseline and end of study assessments.
  RMSSD is a measurement of Heart Rate Variability, measured in milliseconds (ms) using electrocardiography.
Difference and change in Standard Deviation Normal RR Intervals (SDNN). | 12 weeks (baseline to 12 weeks)
  1. Difference in SDNN between COVID and non-COVID participants at rest on baseline assessment.
  2. Change in SDNN between COVID intervention and COVID usual care group at rest on baseline and end of study assessments.
  SDNN is a measurement of Heart Rate Variability, measured in milliseconds (ms) using electrocardiography.
Difference and change in low-frequency power (LF). | 12 weeks (baseline to 12 weeks)
  1. Difference in LF between COVID and non-COVID participants at rest on baseline assessment.
  2. Change in LF between COVID intervention and COVID usual care group at rest on baseline and end of study assessments.
  LF (absolute power) is a measurement of Heart Rate Variability, measured in milliseconds squared (ms2) using electrocardiography.
Difference and change in high-frequency power (HF). | 12 weeks (baseline to 12 weeks)
  1. Difference in HF between COVID and non-COVID participants at rest on baseline assessment.
  2. Change in HF between COVID intervention and COVID usual care group at rest on baseline and end of study assessments.
  HF (absolute power) is a measurement of Heart Rate Variability, measured in milliseconds squared (ms2) using electrocardiography.
Difference and change in low-frequency power (LFnu). | 12 weeks (baseline to 12 weeks)
  1. Difference in LFnu between COVID and non-COVID participants at rest on baseline assessment.
  2. Change in LFnu between COVID intervention and COVID usual care group at rest on baseline and end of study assessments.
  LFnu (relative power) is a measurement of Heart Rate Variability, measured in normal units using electrocardiography.
Difference and change in low-frequency power (HFnu). | 12 weeks (baseline to 12 weeks)
  1. Difference in HFnu between COVID and non-COVID participants at rest on baseline assessment.
  2. Change in HFnu between COVID intervention and COVID usual care group at rest on baseline and end of study assessments.
  HFnu (relative power) is a measurement of Heart Rate Variability, measured in normal units using electrocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Coventry University, Coventry, West Midlands, United Kingdom

REFERENCES:
- [Derived] Rahman M, Russell SL, Okwose NC, Hood OMA, Harwood AE, McGregor G, Raleigh SM, Sandhu H, Roden LC, Maddock H, Banerjee P, Jakovljevic DG. Cardiovascular implications and physical activity in middle-aged and older adults with a history of COVID-19 (CV COVID): a protocol for a randomised controlled trial. Trials. 2023 May 13;24(1):328. doi: 10.1186/s13063-023-07360-7. PMID 37179415